CLINICAL TRIAL: NCT02093234
Title: Changing the Healthcare Delivery Model:A Community Health Worker/Mobile Chronic Care Team Strategy
Brief Title: Changing the Healthcare Delivery Model
Acronym: C4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PCORI- IH-1304-6797; IH-1304-6797 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2016-09

CONDITIONS: Diabetes Type 2
Keywords: self care of diabetes type 2 patients; mobile health cell phone application impact on health; community health workers impact on health
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Navigation; Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobile health care application (Active Comparator): Patients will be assisted with managing their health by a cell phone application used to promote self care for patients with diabetes.
  Interventions: Behavioral: mobile health care application
- Community Health Worker (CHW) (Active Comparator): CHWs assist study patients in managing there health care in various ways.
  Interventions: Behavioral: Community Health Worker (CHW)
- CHWs and mobile health care application (Experimental): Patients will receive assistance in managing their health from both CHWs and the mobile health cell phone application
  Interventions: Behavioral: CHWs and mobile health care application

INTERVENTIONS:
Behavioral: mobile health care application — mobile health application for cell phones to assist patients in managing their diabetes.
  Other Names: Care 4 Life
  Arms: Mobile health care application
Behavioral: CHWs and mobile health care application — CHWs will assist diabetic patients in managing their health in conjunction with the mobile health care application.
  Other Names: Care 4 Life and patient navigators
  Arms: CHWs and mobile health care application
Behavioral: Community Health Worker (CHW) — CHWs assist patients in managing their diabetes in various ways.
  Other Names: Patient navigators
  Arms: Community Health Worker (CHW)

SUMMARY:
This is a randomized controlled trial comparing 3 strategies to improve wellness behaviors and clinical goals for diabetes type 2(DM2) Medicaid patients. A patient interactive cell phone disease management system plus a community health worker (CHW) is superior to either a cell phone system or a CHW alone to activate DM2 Medicaid patients to improve a composite of 7 Wellness Behaviors and 6 Clinical Goals.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing 3 strategies to improve wellness behaviors and clinical goals for DM2 Medicaid patients with uncontrolled DM.

* Group 1 will be assisted by the Voxiva Care4Life mobile health disease management program (C4L) provided on the patient's cell phone.
* Group 2 will be assisted by CHWs who are members of the outpatient medical home health team.
* Group 3 will be assisted by both the Voxiva Care4Life mHealth disease management system (C4L) and a CHW.

Hypotheses:

1. A patient interactive cell phone disease management system plus a community health worker (CHW) is superior to either a cell phone system or a CHW alone to activate DM2 Medicaid patients to improve a composite of 7 Wellness Behaviors and 6 Clinical Goals.
2. A patient interactive cell phone disease management system will activate Medicaid patients with type 2 diabetes (DM2) to improve the composite of 7 wellness behaviors and 6 clinical outcomes by 25% or greater compared to baseline

Expected Outcomes:

Primary outcomes:

1. Superior improvement over baseline of the composite of Wellness Behaviors and Clinical Outcomes in the CHW plus C4L group compared to the CHW alone and cell phone alone groups.
2. Improvement by 25% or greater over baseline of the composite of Wellness Behaviors and Clinical Outcomes for patients using C4L alone.

Secondary outcomes:

Improvement in both clinical and behavior endpoints. Endpoints to be compared across the three treatment arms include:

1. mean HbA1c,
2. mean LDLc Cholesterol
3. average BP if hypertensive
4. Patient distress measured with Fisher Brief Diabetes Distress Screening Instrument

4) Medication adherence measured with Morisky Medication Adherence Survey 5) Healthcare utilization: ER, acute clinic visits, hospitalizations

Anticipated results and impact on healthcare:

Mobile health has great potential to enhance DM2 patient health behaviors and clinical outcomes both alone and, even better, with assistance of a CHW. mHealth systems can be provided to a wide range of urban and rural DM2 patients resulting in an affordable, a more efficient patient-driven/centered health delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years old
* Medicaid insurance coverage, Medicare insurance coverage or Affordable Health Care Act insurance coverage
* Fluent in English or Spanish and able to read a text message
* Diagnosed with diabetes mellitus type 2 and A1C is > 8%

Acceptable values will be either :

* A1c obtained within one month prior to baseline (as long as there were no diabetes changes made during that month) or
* A new A1c measured at the baseline screening visit.
* Meets < 10 of the wellness behaviors and clinical goals if diagnosed with hypertension Meets < 9 of the wellness behaviors and clinical goals if not diagnosed with hypertension

Exclusion Criteria:

* Stage 5 chronic kidney disease or end stage renal disease on dialysis
* Terminal illness (expected survival of less than one year)
* Severe dementia or uncontrolled mental illness
* Gestational diabetes mellitus
* Use of an insulin pump
* Inability to use a cellular phone
* Unable to use software application on cellular phone
* Pregnant or planning to get pregnant

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Katz, MD, Principal Investigator — Medical Faculty Assoc. Inc, GWUniv
Locations (1):
- Medical Faculty Assoc Inc, GWUniv, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcomes measures will be made available with 6 months of study completion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 medical clinic sites in Washington DC. Each site had its' own Principal Investigator ,research coordinator and community health worker. Recruitment started April 2014 and ended July 2015. The study period for each participant was 1 year.
Period: Overall Study
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Started | 56 | 56 | 54
Completed | 53 | 52 | 50
Not Completed | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application | Total
Number analyzed (Participants) | 56 | 56 | 54 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (1.51) | 53.3 (1.21) | 53.2 (1.25) | 52.9 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 41 | 120
  Male | 19 | 14 | 13 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 51 | 51 | 49 | 151
  Other race | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Unmet Behaviors/Goals That Were Not Achieved at Year 1
Description: The study staff will determine the status of the 13 behaviors/goals for the year prior to study enrollment. Our primary endpoint will be the mean change after 1 year in number of behaviors/goals met from baseline.
Time Frame: baseline and 1 year
Population: Sample size estimates were based on the study hypotheses and the associated primary endpoint. Dropouts were analyzed using intention to treat methodology.
Measure: Mean (Standard Error); unit: incomplete behaviors/goals
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Number analyzed (Participants) | 56 | 56 | 54
incomplete behaviors/goals | -1.5 (0.17) | -1.7 (0.29) | -1.1 (0.29)
Statistical Analysis 1: Comparison: Mobile Health Care Application vs Community Health Worker (CHW) vs CHWs and Mobile Health Care Application; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Change in Distress From Baseline as Measured With Fisher Brief Diabetes Distress Screening Instrument
Description: Participants completed the Fisher Brief Diabetes Screening Instrument at baseline and after 1 year of intervention. The instrument consists of 4 questions regarding how participants feel about dealing with diabetes. They are answered using a scale that goes from 1-6, 1= not a bother and 6=very bothersome. Range 4-24.
  Low distress < 12 : moderate / high distress > or = 12.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Number analyzed (Participants) | 56 | 56 | 54
units on a scale | -3.5 (0.71) | -3.7 (1.1) | -4.4 (0.89)
Statistical Analysis 1: Comparison: Mobile Health Care Application vs Community Health Worker (CHW) vs CHWs and Mobile Health Care Application; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Secondary Outcome: Change in Hemoglobin A1C
Description: Change in HbA1c after 1 year from baseline
Time Frame: Baseline and 1 year
Measure: Mean (Standard Error); unit: Percentage of total hemoglobin
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Number analyzed (Participants) | 56 | 56 | 54
Percentage of total hemoglobin | -1.3 (0.20) | -1.2 (0.38) | -1.2 (0.37)
Statistical Analysis 1: Comparison: Mobile Health Care Application vs Community Health Worker (CHW) vs CHWs and Mobile Health Care Application; Test type: Superiority or Other; p < 0.0001, Chi-squared

4. Secondary Outcome: Change in Medication Adherence
Description: Medication adherence Improvement from baseline after 1 year as measured by the Morisky Medication Adherence Survey. Range 1-4 . 1= least adherent , 4= most adherent
Time Frame: baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Number analyzed (Participants) | 53 | 52 | 50
units on a scale | 0.4 (0.19) | 0.09 (0.24) | 0.3 (0.31)
Statistical Analysis 1: Comparison: Mobile Health Care Application vs Community Health Worker (CHW) vs CHWs and Mobile Health Care Application; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected.
Description: Adverse event data was not collected due to the type of intervention used in this trial. The intervention was not a drug , biological product or device that is subject to FDA regulation.
Arm/Group | Mobile Health Care Application | Community Health Worker (CHW) | CHWs and Mobile Health Care Application
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will conduct a peer review of the research report before it may be published.